CLINICAL TRIAL: NCT03932851
Title: Clinical Study on the Effect of IVF-ET on Mother-to-child Transmission of Hepatitis B Virus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wei Yi, Director, Head of Obstetrics and Gynecology, Beijing Ditan Hospital
Other Study IDs: KY2018-012
Record Dates: First submitted 2019-04-15; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBsAg(+) pregnant woman: Data from pregnant women during pregnancy (including age, maternal history, liver function during pregnancy, HBV DNA in early pregnancy and before delivery, comorbidities and complications during pregnancy, antiviral use before and during pregnancy, and HBV infection status in fathers) Newborn birth data (including body length, weight, Apgar score, feeding status, hepatitis B vaccination, hepatitis B immunoglobulin use, HBsAg at birth and 7 months after birth, HBV DNA). The newborns born to HBV-infected pregnant women were divided into HBV DNA-negative group, low-viral group, and high-viral group according to HBV DNA status. The HBV infection status of these newborns was counted in July, and the different viral loads were tested. The impact of HBV mother-to-child transmission.
  Interventions: Other: IVF-ET
- HBsAg(-) pregnant woman: Data from pregnant women during pregnancy (including age, maternal history, liver function during pregnancy, HBV DNA in early pregnancy and before delivery, comorbidities and complications during pregnancy, antiviral use before and during pregnancy, and HBV infection status in fathers) Newborn birth data (including body length, weight, Apgar score, feeding status, hepatitis B vaccination, hepatitis B immunoglobulin use, HBsAg at birth and 7 months after birth, HBV DNA).
  Interventions: Other: IVF-ET

INTERVENTIONS:
Other: IVF-ET — HBV-infected pregnant women and non-HBV-infected pregnant women underwent IVF operation

SUMMARY:
This study is intended to retrospectively collect HBV-infected pregnant women and non-HBV-infected pregnant women who have been born in IVF in the investigators' hospital, collect pregnant women's data during pregnancy, newborn birth data, and hepatitis B virus in July after birth of newborns born to HBV-infected pregnant women. Infection, explore the impact of HBV infection on IVF outcomes and whether IVF operations increase the risk of mother-to-child transmission of HBV.

DETAILED DESCRIPTION:
This study is a retrospective study that only retrospectively collects a variety of patient data and does not perform any treatment or examination on the patient. The research design is as follows: 1. All patients with HBV-infected pregnant women and non-HBV-infected pregnant women who had undergone IVF operation were retrospectively collected from the investigators' hospital HIS system. 2.Collecting pregnant women's data from the HIS system (including age, maternal history, liver function during pregnancy, HBV DNA in early pregnancy and before delivery, complication and complications during pregnancy, antiviral use before and during pregnancy, father HBV infection Status), neonatal birth data (including body length, weight, Apgar score, feeding status, hepatitis B vaccination, hepatitis B immunoglobulin use, HBsAg at birth and 7 months after birth, HBV DNA). 3. Statistical analysis: (1) Compare the body length, body weight, Apgar score of newborns born to pregnant women with HBV infection and non-HBV infection, and understand the effect of HBV infection on IVF outcomes. (2) Newborns born to HBV-infected pregnant women were divided into HBV DNA-negative group, low-viral group, and high-viral group according to HBV DNA status. The HBV infection status of these newborns was counted in July, and the different viral loads were tested. The impact on mother-to-child transmission of HBV. (3) When discussing whether IVF operation increases the rate of mother-to-child transmission of HBV, it is more scientific and persuasive to use HBV-infected pregnant women who have not been operated with IVF, but the incidence of twins in IVF is significantly higher than that of natural pregnancy. Further lead to premature birth, postpartum hemorrhage, cesarean section rate, etc., the weight and length of newborns are also affected, so it is difficult to match the appropriate population, so this study decided to HBV infection rate of different HBV DNA load IVF Compared with the literature, the corresponding viral load of HBV infection was compared with the rate of mother-to-child transmission of IVF pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who have been IVF-operated
* HBV-infected pregnant women need to be positive for HBsAg for more than half a year.

Exclusion Criteria:

* Combined with pregnancy-induced hypertension, premature rupture of membranes, prenatal bleeding and other diseases;
* history of amniocentesis during pregnancy;
* combined with other viral infections: such as HCV, HIV, CMV.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All enrolled subjects are pregnant women
Study Population: All HBV-infected pregnant women who have been IVF-operated and non-HBV-infected pregnant women, HBV-infected pregnant women need to be positive for HBsAg for more than half a year.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Maternal and infant block failure rate in newborns | up to 28 weeks
  Maternal and infant block failure rate in newborns

SECONDARY OUTCOMES:
The length of the newborn and the incidence of various complications during pregnancy. | up to 28 weeks
  The length, weight, Apgar score of the newborn and the incidence of various complications during pregnancy.
The weight of the newborn and the incidence of various complications during pregnancy. | up to 28 weeks
  The weight of the newborn and the incidence of various complications during pregnancy.
The Apgar score of the newborn and the incidence of various complications during pregnancy. | up to 28 weeks
  The Apgar score of the newborn and the incidence of various complications during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Pregnant women, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided